CLINICAL TRIAL: NCT04245397
Title: A Phase 1, Open-Label, Dose-Escalation With Expansion Study of SX-682 Alone and in Combination With Oral or Intravenous Decitabine in Subjects With Myelodysplastic Syndrome
Brief Title: Study of SX-682 Alone and in Combination With Oral or Intravenous Decitabine in Subjects With Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Syntrix Biosystems, Inc. (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); AdventHealth (Other); Emory University (Other); University of Miami (Other); Mayo Clinic (Other); Montefiore Medical Center (Other); National Cancer Institute (NCI) (NIH); Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SX682-MDS-102; R44HL142389 (NIH); R44CA291622 (NIH)
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndromes
Keywords: Immunotherapy; Chemokine receptor blockade; Myeloid-derived supressor cells
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Intervention Model Description: In this sequential model initially participant groups will enroll to receive SX-682 for six 28 day cycles in a dose escalation phase. A 3 + 3 participant design will be used to determine the safe dose. After 6 cycles at the specified dose of SX-682, SX-682 treatment can be continued. Once the safe dose level of SX-682 is determined, then participants will be enrolled at the this safe dose level of SX-682 in an expansion phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation of SX-682 (Experimental): Escalating oral doses of SX-682 (study drug) of 25, 50, 100, 200 and 400 mg twice-daily (i.e., 50, 100, 200, 400 and 800 mg total each day.
  Interventions: Drug: SX-682
- Expansion of SX-682 alone (lower risk patients, naive to hypomethylating agents) (Experimental): Expansion of oral doses of SX-682 (study drug) at 200 mg twice daily (recommended phase 2 dose) in lower risk patients who have never received hypomethylating agents.
  Interventions: Drug: SX-682
- Expansion of SX-682 alone (lower risk patients, failed on hypomethylating agents) (Experimental): Expansion of oral doses of SX-682 (study drug) at 200 mg twice daily (recommended phase 2 dose) in lower risk patients who failed on hypomethylating agents.
  Interventions: Drug: SX-682
- Expansion of SX-682 with decitabine (lower risk patients, naive to hypomethylating agents) (Experimental): Expansion of oral doses of SX-682 (study drug) at 100 mg twice daily with decitabine in lower risk patients who have never received hypomethylating agents.
  Interventions: Drug: SX-682; Drug: Decitabine
- Expansion of SX-682 with decitabine (lower risk patients, failed on hypomethylating agents) (Experimental): Expansion of oral doses of SX-682 (study drug) at 100 mg twice daily with decitabine in lower risk patients who failed on hypomethylating agents.
  Interventions: Drug: SX-682; Drug: Decitabine
- Expansion of SX-682 alone (higher risk patients, failed on hypomethylating agents) (Experimental): Expansion of oral doses of SX-682 (study drug) at 200 mg twice daily (recommended phase 2 dose) in higher risk patients who failed on hypomethylating agents.
  Interventions: Drug: SX-682
- Expansion of SX-682 with decitabine (higher risk patients, naive to hypomethylating agents) (Experimental): Expansion of oral doses of SX-682 (study drug) at 100 mg twice daily with decitabine in higher risk patients who have never received hypomethylating agents.
  Interventions: Drug: SX-682; Drug: Decitabine
- Expansion of SX-682 with decitabine (higher risk patients, failed on hypomethylating agents) (Experimental): Expansion of oral doses of SX-682 (study drug) at 100 mg twice daily with decitabine in higher risk patients who failed on hypomethylating agents.
  Interventions: Drug: SX-682; Drug: Decitabine

INTERVENTIONS:
Drug: SX-682 — SX-682 is an oral small molecule selective inhibitor of C-X-C Motif Chemokine Receptor 1 (CXCR1) and CX-C Motif Chemokine Receptor 2 (CXCR2)
Drug: Decitabine — Decitabine is a hypomethylating agent.
  Other Names: DEC-C
  Arms: Expansion of SX-682 with decitabine (higher risk patients, failed on hypomethylating agents); Expansion of SX-682 with decitabine (higher risk patients, naive to hypomethylating agents); Expansion of SX-682 with decitabine (lower risk patients, failed on hypomethylating agents); Expansion of SX-682 with decitabine (lower risk patients, naive to hypomethylating agents)

SUMMARY:
This study will determine the safety profile, maximum tolerated dose (MTD), dose-limiting toxicities (DLT), and recommended Phase 2 dose (RP2D) of SX-682 in the treatment of patients with Myelodysplastic Syndromes (MDS).

DETAILED DESCRIPTION:
Participants will receive twice daily oral SX-682 for six 28 day cycles. If patients are responding well to the treatment they can continue SX-682 treatment. The first participants will be administered 25 mg orally twice daily. Unless dose limiting toxicities occur, participants will enroll and receive the following increasing twice daily doses of SX-682: 50 mg, 100 mg, 200 mg, and 400 mg.

After establishing the maximum tolerated dose 140 additional participants will be enrolled at the recommended phase 2 dose. Participants will receive continuous SX-682 twice daily oral therapy in 28-day cycles for a total of 6 cycles. The expansion dose cohort will be stratified into IPSS (a) low and intermediate-1 (N=20 SX-682 alone in HMA naive, N=20 SX-682 alone in HMA failure, N=20 SX-682 + DEC-C in HMA-naïve, N=20 SX-682 + DEC-C in HMA-failure) and (b) intermediate-2 and high risk (N=20 SX-682 alone in HMA failure, N=20 SX-682 + DEC-C in HMA-naive, N=20 SX-682 + DEC-C in HMA-failure) MDS. For patients responding well at the end of 6 cycles treatment may continue until disease progression or an adverse event leads to SX-682 discontinuation. Except for blood product transfusions, concurrent therapy for Myelodysplastic Syndromes is not permitted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS by World Health Organization criteria, and either

  1. International Prognostic Scoring System (IPSS) low risk or intermediate-1 risk patients without 5q deletion:

     i. Dose escalation portion: failed prior treatment with at least 4 cycles started of a hypomethylating agent (HMA; azacitidine or decitabine) defined as no response to treatment, loss of response at any time point, or progressive disease/intolerance to therapy.

     ii. Dose expansion portion: failed prior treatment defined as no response to treatment with at least 4 cycles started of HMA, loss of response at any time point, or progressive disease/intolerance to therapy ("HMA failure"); or no prior treatment with HMA ("HMA naive").
  2. IPSS low risk or intermediate-1 risk patients with 5q deletion:

     i. Dose escalation portion: failed prior treatment with at least 4 cycles started of lenalidomide and 4 cycles of hypomethylating agent (azacitidine or decitabine) defined as no response to treatment, loss of response at any time point, or progressive disease/intolerance to therapy.

     ii. Dose expansion portion: same as non-del(5q) lower risk cohort + requirement of failed prior treatment with lenalidomide defined as no response to treatment with at least 4 cycles started of lenalidomide, loss of response at any time point, or progressive disease/intolerance to therapy.
  3. IPSS intermediate-2 risk or high risk patients: HMA failure or HMA naïve as defined above.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Screening laboratory values:

  1. Renal glomerular filtration rate (GFR) ≥ 30 ml/min;
  2. Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) ≤ 3.0 times upper limit of normal;
  3. Bilirubin < 1.5 times upper limit of normal;
  4. No history of HIV being HIV positive;
  5. No active Hepatitis B or Hepatitis C infection.
* Life expectancy ≥ 12 weeks.
* Women of childbearing potential (WOCBP) must use study specified contraception.
* WOCBP demonstrate negative pregnancy test.
* Not breastfeeding.
* Men sexually active must use study specified contraception.

Exclusion Criteria:

* Use of chemotherapeutic agents or experimental agents for MDS within 14 days of the first day of study drug treatment.
* Use of erythroid stimulating agents, Granulocyte-colony stimulating factor (G-CSF), or Granulocyte-macrophage colony-stimulating factor (GM-CSF) within 14 days of the first day of study drug treatment, or during the study.
* Mean triplicate heart rate-corrected QT interval (QTc) > 500 msec.
* Any of the following cardiac abnormalities:

  1. QT interval > 480 msec corrected using Fridericia's formula;
  2. Risk factors for Torsade de Pointes;
  3. Use of medication that prolongs the QT interval with the exception of drugs that are considered absolutely essential for the care of the subject;
  4. Myocardial infarction ≤ 6 months prior to first day of study drug treatment;
  5. Unstable angina pectoris or serious uncontrolled cardiac arrhythmia.
* Any serious or uncontrolled medical disorder.
* Prior malignancy within the previous 2 years except for local cancers that have been cured; or patients who have been adequately treated and have low risk of reoccurrence.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Use of other investigational drugs within 30 days of study drug administration.
* Major surgery within 4 weeks of study drug administration.
* Live-virus vaccination within 30 days of study drug administration.
* Allergy to study drug component.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
SX-682 Maximum Tolerated Dose (MTD) | Up to 28 days in the 28 day Cycle 1.
  Participants cohorts will be enrolled at increasing doses of SX-682. The highest SX-682 dose tested at which no more than 1 of 6 participants experiences a dose limiting toxicity will define the SX-682 MTD
SX-682 Dose Limiting Toxicities (DLT) | Up to 28 days in the 28 day Cycle 1.
  Number of participants experiencing DLTs.

SECONDARY OUTCOMES:
Participants Experiencing a Treatment Response | At the end of Cycle 6 (each cycle is 28 days).
  The percentage of participants experiencing a complete remission, partial remission, or stable disease according to the International Working Group Response Criteria.
SX-682 Delayed Dose Limiting Toxicities | From the beginning of Cycle 2 to the end of Cycle 6 (each cycle is 28 days).
  Number of delayed DLTs experienced by participants.
Adverse Events | At the end of Cycle 6 (each cycle is 28 days).
  Number of participants experiencing adverse events (AEs).
SX-682 Single Dose Maximum Plasma Concentration (Cmax) | Day 1 of Cycle 1 (each cycle is 28 days).
  Blood samples will be collected before and after the first dose of SX-682 on Day 1 of Cycle 1.
SX-682 Steady-State Maximum Plasma Concentration (Css max) | Day 15 of Cycle 1 (each cycle is 28 days).
  Blood samples will be collected before and after the first dose of SX-682 on Day 15 of Cycle 1.
SX-682 Steady-State Minimum Plasma Concentration (Css min) | Day 15 of Cycle 1 (each cycle is 28 days).
  Blood samples will be collected before and after the first dose of SX-682 on Day 15 of Cycle 1.

CONTACTS AND LOCATIONS:
Overall Officials: David A Sallman, MD, Principal Investigator — Moffitt Cancer Center
Locations (7):
- United States (7):
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - AdventHealth Medical Group & Bone Marrow Transplant at Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No